CLINICAL TRIAL: NCT06880770
Title: Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Plozasiran in Adults With Severe Hypertriglyceridemia at High Risk of Acute Pancreatitis (SHASTA-5 Study)
Brief Title: Study of Plozasiran in Adults With Severe Hypertriglyceridemia at Risk of Acute Pancreatitis
Acronym: SHASTA-5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-3011
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — plozasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plozasiran Injection (Experimental): Plozasiran by SC injection every 3 months (Q3M) through completion of the randomized period
  Plozasiran by SC injection Q3M through completion of the OLE period
  Interventions: Drug: Plozasiran
- Placebo (Experimental): calculated volume to match active treatment by SC injection (randomized period)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plozasiran — ARO-APOC3 injection
  Other Names: ARO-APOC3
  Arms: Plozasiran Injection
Drug: Placebo — sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of plozasiran in approximately 288 adult participants with severe hypertriglyceridemia (SHTG) and history of at least two prior acute pancreatitis (AP) events not attributed to other etiologies, with at least one occurring within the last 12 months prior to screening. Eligible participants will be randomly assigned in a double-blind manner to either receive plozasiran 25 mg by subcutaneous (SC) injection every three months (Q3M) or matching placebo. Enrolled participants will be counseled to remain on the specified low-fat diet and background medications throughout the study. Following completion of the double-blind treatment period, or if the participant has a positively adjudicated AP event (whichever occurs first), participants will transition to the 12-month Open-Label Extension (OLE) treatment period receiving plozasiran 25 mg by SC injection Q3M.

ELIGIBILITY:
Inclusion Criteria:

* Males, or nonpregnant (who do not plan to become pregnant) nonlactating females
* Established diagnosis of SHTG and prior documented evidence of fasting TG levels of ≥ 880 mg/dL (≥ 10 mmol/L)
* Documented evidence of at least 1 prior AP event not attributed to other etiologies occurring within the last 60 months prior to Screening.
* Fasting low-density lipoprotein cholesterol (LDL-C) ≤ 130 mg/dL (≤ 3.37 mmol/L) at Screening
* Screening hemoglobin A1c (HbA1c) ≤ 9.5%
* Willing to follow diet counseling and maintain a stable low-fat diet
* Must be on standard of care lipid and TG-lowering medications per local guidelines (unless documented as intolerant, or a treatment failure as determined by the Investigator)

Exclusion Criteria:

* Use of any hepatocyte-targeted small interfering ribonucleic acid (siRNA) that targets lipids and/or triglycerides within 365 days before Day 1, except inclisiran.
* Use of any other hepatocyte targeted siRNA or antisense oligonucleotide molecule within 60 days or within 5 half-lives lives before day 1. Whichever is longer.
* AP ≤ 4 weeks prior to Randomization/Day 1
* Body mass index (BMI) > 45 kg/m^2
* Any planned bariatric surgery or similar procedures to induce weight lost starting at consent through End of Study (EOS)
* Planned coronary intervention (e.g. stent placement or heart bypass) during the study
* History of arterial revascularization within 16 weeks of Screening
* History of acute coronary syndrome event within 24 weeks of Screening
* Recent atherosclerotic cardiovascular disease (ASCVD) event within 24 weeks of Screening
* Recent unstable or symptomatic cardiac arrhythmia (including any associated medication changes) within 90 days of Screening. Individuals with stable well-controlled atrial arrhythmia will be allowed to participate in the study
* History of pacemaker or automatic implantable cardioverter defibrillators implant within 30 days before Screening
* New York Heart Association Class III-IV heart failure or last known ejection fraction of < 30%
* Current diagnosis of nephrotic syndrome
* Chronic kidney disease, defined by an estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73 m^2
* Liver disease defined as cirrhosis or Child-Pugh Class B and C, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5× Upper Limit of Normal (ULN) at Screening

Note: Additional Inclusion/Exclusion Criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Positively Adjudicated AP Event (Event Occurring More Than 10 Days After First Dose of Study Drug) | Randomization up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)]

SECONDARY OUTCOMES:
Percent Change from Baseline in Fasting Serum Triglyceride (TG) Levels | Baseline up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)
Proportion of Participants Who Achieve Average Fasting TG Levels of < 880 mg/dL (10 mmol/L) | From Month 3 up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)
Proportion of Participants Who Achieve Fasting TG Levels of < 500 mg/dL (5.65 mmol/L) | From Month 3 up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)
Time to First Occurrence of Major Abdominal Pain Event (Event Occurring More Than 10 Days After the First Dose of Study Drug). | Randomization up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)
Change from Baseline in Patient-Reported Productivity and Activity Impairment as Assessed by the Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP) Score | Baseline up to end of Double Blind Treatment Period Study compared to placebo (Approximate Maximum 50 Months)
Change from Baseline in Patient-Reported Health Status as Assessed by the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Score | Baseline up to end of Double Blind Treatment Period compared to placebo (Approximate Maximum 50 Months)
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) compared to placebo | From first dose of study drug up to Study Completion (Approximate Maximum 62 Months)
Rate of Occurrence of Adjudicated Major Cardiovascular Events (MACE) | From first dose of study drug up to Study Completion (Approximate Maximum 62 Months)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (12):
  - Research Site, Los Angeles, California
  - Clinical Research Site 4, Santa Clarita, California
  - Clinical Research Site 6, Springfield, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, St Louis, Missouri
  - Clinical Research Site 5, North Platte, Nebraska
  - Clinical Research Site 3, Greensboro, North Carolina
  - Research Site, Wilmington, North Carolina
  - Clinical Research Site 7, Philadelphia, Pennsylvania
  - Clinical Research Site 1, Mesquite, Texas
  - Clinical Research Site 2, San Antonio, Texas
- Research Site, Graz, Austria
- Brazil (4):
  - Research Site, Fortaleza, Ceará
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Pôrto Alegre, Rio Grande do Sul
- Bulgaria (7):
  - Research Site, Burgas
  - Research Site, Pleven
  - Research Center, Plovdiv
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
- China (11):
  - Research Center, Beijing, Beijing Municipality
  - Research Site, Guiyang, Guizhou
  - Research Site, Harbin, Heilongjiang
  - Research Center, Baotou, Inner Mongolia
  - Research Site, Chifeng, Inner Mongolia
  - Research Center, Nanchang, Jiangxi
  - Research Center, Shanghai, Shanghai Municipality
  - Research Center, Hangzhou, Zhejiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Nanjing
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Szeged
- Jordan (3):
  - Research Site, Amman
  - Research Center, Amman
  - Research Center, Irbid
- Research Site, Muscat, Oman
- Serbia (4):
  - Research Center, Belgrade
  - Research Site, Belgrade
  - Research Site, Pančevo
  - Research Center, Zaječar
- South Korea (4):
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Busan
  - Research Site, Sejong
  - Research Site, Seoul
- Sweden (2):
  - Research Center, Gothenburg
  - Research Center, Stockholm
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City

IPD SHARING:
Plan to Share IPD: No